CLINICAL TRIAL: NCT00005601
Title: A Phase II Trial of Cisplatinum, Cytosine Arabinoside, Dexamethasone (DHAP) With Rituxan in Patients With Relapsed CD20+ B-Cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy Plus Rituximab in Treating Patients With Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9981; NCI-2012-02326 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000067714 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cisplatin; Cytarabine; Dexamethasone; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab+dexamethasone+cisplatin+cytarabine+sargramostim (Experimental): Patients receive rituximab IV on days 1, 8, 15, and 22 for the first course only. Patients receive dexamethasone orally or IV on days 1-4, cisplatin IV continuously for 24 hours on day 1, cytarabine IV over 3 hours every 12 hours for 2 doses on day 2, and sargramostim (GM-CSF) subcutaneously on days 3-12 or until blood counts recover. Chemotherapy repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.
  Interventions: Biological: rituximab; Drug: cisplatin; Drug: cytarabine; Drug: dexamethasone; Drug: sargramostim

INTERVENTIONS:
Biological: rituximab
Drug: cisplatin
Drug: cytarabine
Drug: dexamethasone
Drug: sargramostim

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining combination chemotherapy with monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus rituximab in treating patients who have relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response rate to cisplatin, cytarabine, and dexamethasone (DHAP) plus rituximab in patients with relapsed CD20+ B-cell non-Hodgkin's lymphoma.
* Determine the percentage of patients able to proceed to transplant after two courses of this treatment regimen.
* Determine the duration of response and overall survival of the patients not proceeding to transplant after two courses of this treatment regimen.

OUTLINE: Patients receive rituximab IV on days 1, 8, 15, and 22 for the first course only. Patients receive dexamethasone orally or IV on days 1-4, cisplatin IV continuously for 24 hours on day 1, cytarabine IV over 3 hours every 12 hours for 2 doses on day 2, and sargramostim (GM-CSF) subcutaneously on days 3-12 or until blood counts recover. Chemotherapy repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 17-50 patients will be accrued for this study within 11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20+ B-cell non-Hodgkin's lymphoma

  * Relapsed following chemotherapy and eligible for platinum-containing regimen
* Measurable disease

  * Must be at least 1.5 x 1.5 cm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 1.5 times upper limit of normal

Cardiovascular:

* No uncontrolled hypertension

Other:

* HIV negative
* No other active malignancy
* No uncontrolled diabetes mellitus
* No uncontrolled peptic ulcer disease
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2000-10; Primary Completion 2003-07 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
response | Up to 5 years

SECONDARY OUTCOMES:
percentage of patients able to proceed to transplant after two courses of this treatment regimen | Up to 5 years
duration of response | Up to 5 years
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Witzig TE, Geyer SM, Kurtin PJ, Colgan JP, Inwards DJ, Micallef IN, LaPlant BR, Michalak JC, Salim M, Dalton RJ, Moore DF Jr, Reeder CB; North Central Cancer Treatment Group. Salvage chemotherapy with rituximab DHAP for relapsed non-Hodgkin lymphoma: a phase II trial in the North Central Cancer Treatment Group. Leuk Lymphoma. 2008 Jun;49(6):1074-80. doi: 10.1080/10428190801993470. PMID 18569634